CLINICAL TRIAL: NCT06799611
Title: An Open, Exploratory Clinical Study to Assess Safety and Efficacy of BCMA-CD3 Bispecific Antibody CM336 in the Treatment of Primary Immune Thrombocytopenia
Brief Title: An Open, Exploratory Clinical Study of CM336 in the Treatment of Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024050
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Immune Thrombocytopenia (ITP); Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention(CM336) (Experimental): CM336 (Anticipated enrollment of 20 to 30 subjects)
  Interventions: Drug: CM336 Injection

INTERVENTIONS:
Drug: CM336 Injection — subcutaneous CM336 administration step-up dosing Dose and frequency of CM336 according to the protocol

SUMMARY:
To evaluate the efficacy and safety of CM336 in the treatment of refractory adult primary immune thrombocytopenia

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for recurrent and refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.

The main pathogenesis of ITP is the loss of platelet autoantigen immune tolerance, which leads to abnormal activation of humoral and cellular immunity. It is characterized by antibody mediated platelet destruction and insufficient platelet production by megakaryocytes. The residual long-term autoreactive plasma cells may be a source of therapeutic resistance to autoimmune cytopenia. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. Therefore, the strategy of simply eliminating B cells may not work, because LLPC will continue to produce pathogenic antibodies. However, targeting LLPC becomes a new strategy to treat autoimmune diseases.

B-cell maturation antigen (BCMA) is mainly restricted in some B-cell subsets and plasma cells, but not in other normal human cells and tissues. BCMA does not maintain normal B-cell homeostasis, but is necessary for long-lived plasma cell survival. Plasma cells are the main antibody-producing cells in the body, and the production of autoantibodies is the main pathogenesis of ITP. BCMA-CD3 bispecific antibody CM336 can bind BCMA-positive B cells and plasma cells, and bind CD3-positive T cells at the same time to induce T cell activation and play the role of T-cell-dependent cellular cytotoxicity (TDCC). CM336 can eliminate BCMA-positive B cells and plasma cells through the above mechanism, directly reduce the production of pathogenic antibodies, and then achieve therapeutic effect. Due to the deep clearance of immune cells by bispecific antibodies, CM336 may achieve the effect of immune reset and cure autoimmune diseases such as ITP. The BCMA-CD3 bispecific antibody teclistamab has been reported to be used in the treatment of refractory systemic lupus erythematosus, systemic sclerosis, primary Sjogren's syndrome, idiopathic inflammatory myopathy, rheumatoid arthritis and other autoimmune diseases, with significant clinical effect and good safety.

Therefore, the investigators designed this clinical trial to evaluate the safety and efficacy of CM336 in the treatment of refractory ITP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above, male or female;
* Conform to the diagnostic criteria of persistent or chronic immune thrombocytopenia (ITP);
* Failure of previous glucocorticoid therapy;
* In the second-line treatment phase, eligible subjects must meet any of the following criteria: (1) Demonstrate no response to treatment with at least one thrombopoietin receptor agonist (including but not limited to recombinant human thrombopoietin [rhTPO], eltrombopag, hetrombopag, avatrombopag, or romiplostim); Fail to achieve sustained response (manifested as non-response, loss of response, or disease relapse) following anti-CD20 monoclonal antibody therapy (e.g., rituximab) or anti-CD38 monoclonal antibody therapy; (2) Exhibit no therapeutic response or experience disease relapse after splenectomy.
* The platelet count was <30×109/L within 48 hours before the first administration;
* ECOG physical state score ≤ 2 points;
* Patients receiving maintenance treatment (including corticosteroids (less than or equal to 20mg prednisone), TPO receptor agonists, etc.) must have a stable dose at least 4 weeks before the first administration;
* Signed and dated written informed consent;

Exclusion Criteria:

* Received any treatment of anti-BCMA antibody drug;
* Accompanied by autoimmune hemolytic anemia, or various secondary and hereditary thrombocytopenia;
* History of any thrombotic or embolic events in the 12 months prior to the first dose or accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage, etc;
* Participated in any other study drug or exposure to other study drugs within 4 weeks or 5 half-lives before the first dose (whichever is longer);
* Use of anticoagulants or any drug with antiplatelet effects (such as aspirin) within 3 weeks before the first dose;
* Treatment with ITP (methylprednisolone, platelet, gamma-globulin infusion or TPO receptor agonist therapy) within 2 weeks before the first dose;
* Splenectomy was performed within 6 months before the first dose;
* Patients who received azathioprine, danazol, cyclosporine A, tacrolimus, sirolimus, etc., within 4 weeks prior to the first dose; or received treatments such as CD20 monoclonal antibodies (e.g., rituximab), CD38 monoclonal antibodies, cyclophosphamide, or vindesine within 3 months prior to the first dose；
* Received a live vaccine within 4 weeks before the first dose, or planned to receive any live vaccine during the clinical trial;
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past;
* Other serious diseases that may limit the subject's participation in this trial (such as diabetes; Hepatic and renal insufficiency; Severe cardiac insufficiency; Myocardial obstruction or unstable arrhythmia or unstable angina pectoris in recent 6 months; Gastric ulcer, etc.);
* Patients with malignant tumors within 5 years before the screening;
* A history of severe recurrent or chronic infection;
* A known or suspected history of immunosuppression, including a history of invasive opportunistic infections;
* Clinically significant laboratory abnormalities at the time of screening;
* HIV antibody or syphilis antibody positive;
* Accompanied by uncontrollable active infection, including hepatitis B, hepatitis C; Pregnant women, suspected pregnancies (positive pregnancy test for human chorionic gonadotropin in urine at screening) and lactating patients;
* Patients with mental disorders who cannot normally obtain informed consent and conduct trials and follow-up;
* Patients whose symptoms of toxicity from pre-trial treatment have not resolved;
* Any other ineligibility for subjects in the study was assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy after CM336 treatment at week 12 | 12 weeks
  Proportion of subjects whose platelet counts ≥ 30×10^9/L and at least two times of baseline platelet count without bleeding at week 12
Safety of CM336 | 52 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after CM336 treatment

SECONDARY OUTCOMES:
Proportion of subjects with a platelet count ≥ 50 × 10^9/L and ≥ 100 × 10^9/L at each visit | 52 weeks
  Proportion of subjects with a platelet count ≥ 50 × 10^9/L and ≥ 100 × 10^9/L at each visit after administration.
Duration from treatment initiation to platelet count ≥30×10^9/L and at least two times of baseline platelet count, platelet count ≥50×10^9/L, platelet count ≥100×10^9/L | 52 weeks
  Duration from treatment initiation to platelet count ≥30×10^9/L and at least two times of baseline platelet count, platelet count ≥50×10^9/L, platelet count ≥100×10^9/L
Cumulative weeks of platelet ≥30×10^9/L and at least two times of baseline platelet count, platelet count ≥50×10^9/L, platelet count ≥100×10^9/L | 52 weeks
  Cumulative weeks of platelet ≥30×10^9/L and at least two times of baseline platelet count, platelet count ≥50×10^9/L, platelet count ≥100×10^9/L
Other efficacy evaluation | 52 weeks
  Platelet counts at each visit
Proportion of subjects receiving emergency treatment | 52 weeks
  Proportion of subjects receiving emergency treatment within 12 weeks and throughout the clinical trial
Changes in world health organization (WHO) bleeding scale | 52 weeks
  Changes in world health organization (WHO) bleeding scale without emergency treatment. Changes of every subject in WHO bleeding score after CM336 treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Measurements of platelet glycoprotein (GP) autoantibodies | 52 weeks
  level of anti-GPIIb/IIIa and Ib/IX antibodies before and after CM336 therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months to 36 months after study completion.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI